CLINICAL TRIAL: NCT00992810
Title: Medial vs. Lateral Approach to Ultrasound-Guided Supraclavicular Block: A Prospective Randomized Controlled Trial
Brief Title: Medial Versus Lateral Approach in Ultrasound (US)-Guided Supraclavicular Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-0451-B
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2010-01

CONDITIONS: Hand or Arm Surgery
Keywords: upper limb; hand; arm; surgery; supraclavicular nerve block; brachial plexus nerve block; ultrasound-guided regional anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lateral-to-Medial Approach (Experimental): Needle approach to the brachial plexus nerves will be made using a lateral-to-medial direction.
  Interventions: Procedure: Lateral-to-Medial Approach
- Medial-to-Lateral Approach (Experimental): Needle approach to the brachial plexus nerves will be made using a lateral-to-medial direction.
  Interventions: Procedure: Media-to-Lateral Approach

INTERVENTIONS:
Procedure: Lateral-to-Medial Approach — Approach of the needle to administer the brachial plexus nerve block will be done in a lateral-to-medial direction.
  Arms: Lateral-to-Medial Approach
Procedure: Media-to-Lateral Approach — Approach of the needle to administer the brachial plexus nerve block will be done in a medial-to-lateral direction.
  Arms: Medial-to-Lateral Approach

SUMMARY:
The ultrasound guided supraclavicular block is a peripheral nerve block which is considered safe, has a fast onset, is dense and provides complete block of the nerves supplying the hand, forearm and arm. However retrospective studies done at Toronto Western Hospital have highlighted the fact that most commonly the ulnar nerve fibres (responsible for sensations in the ring finger, little finger and the corresponding part of hand), sometimes escape this block and need additional supplementary block at a distal peripheral nerve site. It is a confusing fact since all nerve fibres are compactly arranged in a sheath at the supraclavicular level. The local anaesthetic agent at this level should be equally distributed among all nerve fibres. The purpose of this study is to compare two different approaches (medial and lateral) adopted by our clinicians to perform this block and to test the effectiveness of each approach for successful ulnar nerve fibre blockade.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients presenting for upper limb surgery, excluding shoulder surgery
* Age 18-80 yrs
* BMI < 35
* ASA I - III
* Consent for the study

Exclusion Criteria:

* Pre-existing sensory or motor neurodeficit.
* Sensitivity to local anaesthetic agents.
* Patients on anticoagulants or antiplatelet medications (Minidose Aspirin is acceptable) with abnormal coagulation profile.
* Compromised pulmonary reserve due to COPD, Kypho-scoliosis or Restricted lung disease.
* Infection or any obvious pathology at the site of block performance
* History of drug abuse.
* Psychiatric disease or any condition that precludes an informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Successful block of the Ulnar nerve (C8,T1) fibres. Sensory block with a score of '1' at 30 minutes (loss of sensation to pin prick) is considered successful. | 1 hour prior to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada